CLINICAL TRIAL: NCT00005755
Title: Community Based Study on Occupational Asthma
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5109; R01HL062633 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2006-01

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To examine the occupations, industries and exposures in the work-place which were associated with a high risk for asthma and other adverse respiratory health effects, with particular emphasis on specific exposures of predominantly female occupations (irritants, detergents and other asthmagens), and of other high risk major occupations which had not been adequately examined.

DETAILED DESCRIPTION:
BACKGROUND:

Respiratory diseases are strongly related with exposure in the workplace. A considerable proportion of adult onset asthma is associated with these exposures. The importance of occupational risk factors for asthma has been underestimated, particularly among women. The occupational asthma study (ECRHS-OA) forms part of a wider international multicentre survey on respiratory health (European Community Respiratory Health Survey-ECRHS). The first phase of the ECRHS was conducted in 1991/92 and examined risk factors for asthma and atopy in subjects aged 20-44 years. The study updated (ECRHS-II), following-up approximately 17,000 young adults from 12 countries (Australia, Belgium, France, Germany, Iceland, Italy, Norway, Spain, Sweden, Switzerland, UK and USA).

The study provided valid and precise estimates on the importance of specific occupations, industries and exposures in relation to asthma incidence and prevalence, similar estimates for other respiratory symptoms and diseases and also for declines in pulmonary function.

DESIGN NARRATIVE:

Longitudinal, community-based, multicenter study. Those subjects who took part in the first occupational asthma study survey were re-contacted in 1999, to determine risk factors for incidence and remission of asthma, other respiratory symptoms, atopy, changes in bronchial responsiveness and lung function. Subjects were asked to perform a forced spirometry, methacholine challenge and to provide blood samples for IgE testing. A questionnaire administrated by trained interviewers was delivered requesting information on respiratory symptoms and diseases, socio-demographic factors, tobacco smoking, complete occupational history since the last survey, environmental exposures, family history, diet, treatment and use of health services. Modular occupational questionnaires were developed for subjects employed as cleaners, homemakers, welders, metal workers, nurses, and subjects exposed to organic dusts in the paper and textile industries.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1999-05; Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manolis Kogevinas — Municipal Institute of Medical Research

REFERENCES:
- [Background] Zock JP, Kogevinas M, Sunyer J, Almar E, Muniozguren N, Payo F, Sanchez JL, Anto JM; Spanish working group of the European Community Respiratory Health Survey. Asthma risk, cleaning activities and use of specific cleaning products among Spanish indoor cleaners. Scand J Work Environ Health. 2001 Feb;27(1):76-81. doi: 10.5271/sjweh.590. PMID 11266151
- [Background] Zock JP, Kogevinas M, Sunyer J, Jarvis D, Toren K, Anto JM; European Community Respiratory Health Survey. Asthma characteristics in cleaning workers, workers in other risk jobs and office workers. Eur Respir J. 2002 Sep;20(3):679-85. doi: 10.1183/09031936.02.00279702. PMID 12358347
- [Background] Zock JP, Cavalle N, Kromhout H, Kennedy SM, Sunyer J, Jaen A, Muniozguren N, Payo F, Almar E, Sanchez JL, Anto JM, Kogevinas M. Evaluation of specific occupational asthma risks in a community-based study with special reference to single and multiple exposures. J Expo Anal Environ Epidemiol. 2004 Sep;14(5):397-403. doi: 10.1038/sj.jea.7500337. PMID 15361899
- [Background] de Vocht F, Zock JP, Kromhout H, Sunyer J, Anto JM, Burney P, Kogevinas M. Comparison of self-reported occupational exposure with a job exposure matrix in an international community-based study on asthma. Am J Ind Med. 2005 May;47(5):434-42. doi: 10.1002/ajim.20154. PMID 15828067